CLINICAL TRIAL: NCT01357356
Title: A Randomized, Double Blind, Placebo Controlled, Parallel Group, Multicenter Study to Investigate the Efficacy and Safety of SER120 Nasal Spray Formulations in Patients With Nocturia
Brief Title: Multicenter Study to Investigate SER120 Nasal Spray Formulations in Patients With Nocturia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Serenity Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPC-SER120-DB3-201101
Record Dates: First submitted 2011-05-18; First posted 2011-05-20 (Estimated); Results first posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2015-11

CONDITIONS: Nocturia
MeSH Terms: conditions — Nocturia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- SER120 (750 ng/day) (Experimental): SER120 (750 ng/day)
  Interventions: Drug: SER120 (750 ng/day)
- SER120 (1000 ng/day) (Experimental): SER120 (1000 ng/day)
  Interventions: Drug: SER120 (1000 ng/day)
- SER120 (1500 ng/day) (Experimental): SER120 (1500 ng/day)
  Interventions: Drug: SER120 (1500 ng/day)
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SER120 (750 ng/day)
  Arms: SER120 (750 ng/day)
Drug: SER120 (1000 ng/day) — SER120 (1000 ng/day)
  Arms: SER120 (1000 ng/day)
Drug: SER120 (1500 ng/day)
  Arms: SER120 (1500 ng/day)
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of SER120 nasal spray formulations in patients with nocturia for a total duration of 14 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male and female 50 years or older
* Nocturia of 6 or more months duration averaging greater than 2 nocturic episode per night

Exclusion Criteria:

* CHF
* Diabetis Insipidus
* Renal Insufficiency
* Hepatic Insufficiency
* Incontinence
* Illness requiring systemic steroids
* Malignancy within the past 5 years
* Sleep Apnea
* Nephrotic Syndrome
* Unexplained Pelvic Mass
* Urinary Bladder Neurological dysfunction
* Urinary Bladder Surgery or Radiotherapy
* Pregnant or Breast Feeding

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Actual)
Dates: Start 2011-05; Primary Completion 2012-10 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Serenity R&D, New City, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- SER120 750 ng: All participants received SER120 750 ng once daily
- SER120 1000 ng: All participants received SER120 1000 ng once daily
- SER120 1500 ng: All participants received SER120 1500 ng once daily
- Placebo: All participants received Placebo once daily
Period: Overall Study
Arm/Group | SER120 750 ng | SER120 1000 ng | SER120 1500 ng | Placebo
Started | 188 | 188 | 186 | 188
Completed | 166 | 163 | 158 | 171
Not Completed | 22 | 25 | 28 | 17

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population
Groups:
- Total: Total of all reporting groups
Arm/Group | SER120 750 ng | SER120 1000 ng | SER120 1500 ng | Placebo | Total
Number analyzed (Participants) | 186 | 183 | 179 | 186 | 734
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (9.1) | 66.1 (8.9) | 66.0 (9.4) | 66.0 (10.1) | 66.1 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 74 | 75 | 74 | 302
  Male | 107 | 109 | 104 | 112 | 432
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 2 | 5 | 6 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 15 | 18 | 20 | 21 | 74
  White | 165 | 163 | 152 | 155 | 635
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 171 | 171 | 160 | 175 | 677
  Canada | 15 | 12 | 19 | 11 | 57

OUTCOME MEASURES:

1. Primary Outcome: Change in # of Mean Nocturic Episodes Per Night
Description: Change was calculated based on the number of mean nocturic episodes per night between baseline through week 12
Time Frame: 12 weeks
Population: Intent to treat population
Measure: Least Squares Mean (Standard Error); unit: nocturic episodes per night
Arm/Group | SER120 750 ng | SER120 1000 ng | SER120 1500 ng | Placebo
Number analyzed (Participants) | 186 | 183 | 179 | 186
nocturic episodes per night | -1.4 (0.07) | -1.4 (0.07) | -1.6 (0.07) | -1.2 (0.07)

2. Primary Outcome: Percent of Participants With 50% or Greater in Reduction of Nocturic Episodes
Description: Percent of participants achieving at least 50% reduction in mean nocturic episode per night during 12 weeks compared to baseline
Time Frame: 12 weeks
Population: Intent to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | SER120 750 ng | SER120 1000 ng | SER120 1500 ng | Placebo
Number analyzed (Participants) | 186 | 183 | 179 | 186
Participants | 77 | 73 | 93 | 61

ADVERSE EVENTS:
Description: Adverse events were collected from the Safety Population, i.e., any patient who had received one dose of study drug and reported an adverse event.
Arm/Group | SER120 750 ng | SER120 1000 ng | SER120 1500 ng | Placebo
Serious Adverse Events (participants affected / at risk) | 2/188 | 3/186 | 5/184 | 6/187
Other Adverse Events (participants affected / at risk) | 18/188 | 15/186 | 21/184 | 19/187
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SER120 750 ng (N=188) | SER120 1000 ng (N=186) | SER120 1500 ng (N=184) | Placebo (N=187)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tongue neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SER120 750 ng (N=188) | SER120 1000 ng (N=186) | SER120 1500 ng (N=184) | Placebo (N=187)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 9 (9) | 11 (11) | 7 (7)
Headache (Nervous system disorders) | 8 (8) | 5 (5) | 2 (2) | 8 (8)
Hypertension (Vascular disorders) | 4 (4) | 1 (1) | 8 (8) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes